CLINICAL TRIAL: NCT03591380
Title: CAMPath and BELimumab for the Induction of Donor Specific Humoral Transplant Tolerance in Sensitized Kidney Transplant Recipients To Improve Long-Term Allograft Survival
Brief Title: CAMPath and BELimumab for Transplant Tolerance in Sensitized Kidney Transplant Recipients
Acronym: CAMPBEL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment complications due to COVID-19
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: GlaxoSmithKline (Industry); American College of Surgeons (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1385; Protocol Version 8/17/2020 (Other: UW Madison); A539742 (Other: UW Madison); SMPH/SURGERY/TRANSPLANT (Other: UW Madison)
Record Dates: First submitted 2018-05-03; First posted 2018-07-19 (Actual); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Kidney Transplantation
Keywords: Donor Specific Antibody; Donors, Living; Allograft Tolerance
MeSH Terms: interventions — belimumab

STUDY DESIGN:
Intervention Model Description: This study is proposed to be an open-label, single-arm, pilot study to test whether the addition of belimumab, to inhibit the B cell survival factor BLyS at the time of kidney transplantation, to standard or care therapy (alemtuzumab and steroid induction with mycophenolic acid and tacrolimus maintenance immunosuppression) will prevent the prevent the generation of de novo DSA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: Belimumab (Experimental): Belimumab 10mg/kg will be administered IV at the following intervals: at the time of transplant (Day 0), then post-transplant at 2, 4, 8, 12, 16, and 20 weeks.
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — Kidney transplant recipients (n=5) will receive standard of care (SOC) therapy consisting of alemtuzumab and steroid induction with mycophenolic acid and tacrolimus maintenance immunosuppression, plus induction and treatment for 6 months with belimumab.
  Other Names: Benlysta

SUMMARY:
The purpose of this research study is to determine whether kidney transplant recipients who receive belimumab (Benlysta®), combined with the standard of care medications for kidney transplant recipients, is safe and effective in helping prevent new donor specific antibodies (DSA) after transplantation. The presence of DSA increases the risk that the kidney transplant recipient's body will reject the new kidney. The investigators are doing this research because it is estimated that greater than 50% of kidney transplant failures are attributed to antibodies produced in the body, that attack the transplanted organ as a foreign object. DSA produced in the body after a kidney transplant, is thought to occur in 20-50% of patients and is associated with a low likelihood that the organ recipient's body will accept the new kidney. A major unmet need in the kidney transplant area are safe and effective therapies to prevent DSA after transplantation.

DETAILED DESCRIPTION:
Accrual Objective: Kidney transplant recipients (n=5) will receive standard of care (SOC) therapy consisting of alemtuzumab and steroid induction with mycophenolic acid and tacrolimus maintenance immunosuppression, plus induction and treatment for 6 months with belimumab.

Study Design: This is an open-label pilot-study to evaluate the safety and efficacy of belimumab plus standard of care in the prevention of de novo donor specific antibody in adult subjects after kidney transplantation.

The investigators will enroll 5 adult, deceased or living donor kidney transplant recipients who are sensitized, evidenced by: Positive sum Donor Specific Antibody (DSA)<1000 MFI and/or Panel of Reactive Antibodies (PRA)>0%. The primary endpoint of this study is de novo DSA production. There are two main reasons for selecting this patient population for the proposed study. 1) Sensitized patients are known to have higher rates of de novo DSA production and 2) Patients with low levels of DSA (sum DSA<1000 MFI) will enable more fidelity in determining the DSA that is produced de novo.

Kidney transplant recipients will receive the standard of care (alemtuzumab and steroid induction with mycophenolic acid and tacrolimus maintenance immunosuppression), plus six months of therapy with belimumab. Belimumab 10 mg/kg will be administered IV for 6 months at the following intervals: Day of transplant (Day 0), and then at Weeks 2, 4, 8, 12, 16, and 20 post-transplant.

Study Duration: Subjects will be treated for 6 months with belimumab and followed for DSA production for 1 year.

Primary Study Objectives: In this proposal the investigators plan to determine (a) whether the addition of belimumab to the standard of care (SOC: alemtuzumab and steroid induction with mycophenolic acid and tacrolimus maintenance immunosuppression) is safe and effective in preventing de novo DSA production at 1, 3, 6, 9, and 12 months post-transplant.

Secondary efficacy endpoints will be 1) graft survival and function as determined by serum creatinine/eGFR and urine protein at 1, 3, 6, 9, and 12 months 2) rates of acute cellular and antibody mediated rejection, at 1, 3, 6, 9, and 12 months.

Primary Outcomes: To determine whether the addition of belimumab to the standard of care (SOC: alemtuzumab and steroid induction with mycophenolic acid and tacrolimus maintenance immunosuppression) is safe and effective in preventing de novo DSA production 1, 3, 6, 9, and 12 months.

Secondary Outcomes: Secondary endpoints will be 1) graft survival and function as determined by serum creatinine/eGFR and urine protein at 1, 3, 6, 9, and 12 months 2) rates of acute cellular and antibody mediated rejection at 1, 3, 6, 9, and 12 months and 3) the nature, frequency, and severity of serious and non-serious adverse events ≥Grade 2 per Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18-60 years of age
* Planned to receive a deceased or living donor kidney transplant
* Sensitized patients: Positive sum DSA <1000, and/or PRA>0%.
* Subjects must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.
* Female subjects must be post-menopausal, surgically sterilized, or she and/or sexual partner must be willing to use an acceptable method of birth control with a <1% failure rate as stated in the product label from time of study consent, during study participation, and for 16 weeks after the last dose of the study agent (i.e., contraceptive subdermal implant of levonorgestrel or etonogestrel, intrauterine device or intrauterine system, combined estrogen and progestogen oral contraceptive, Injectable progestogen, contraceptive vaginal ring, percutaneous contraceptive patches, or abstinence) for the duration of the study. Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject. The documentation of male sterility can come from the site personnel's: review of subject's medical records, medical examination and/or semen analysis, or medical history interview provided by her or her partner. Note: Mycophenolate mofetil (MMF) affects the metabolism of oral contraceptives and may reduce their effectiveness. As such, women receiving MMF who are using oral contraceptives for birth control should employ an additional method (e.g., barrier method). Mycophenolate can cause fetal harm when administered to a pregnant female. Use of mycophenolate during pregnancy is associated with an increased risk of first trimester pregnancy loss and an increased risk of congenital malformations. Mycophenolate affects the metabolism of oral contraceptives and may reduce their effectiveness. As such, women receiving MMF who are using oral contraceptives for birth control should employ an additional method (e.g., barrier method) resulting in two reliable forms of contraception being used simultaneously before starting study treatments, during therapy, and for 6 weeks after stopping therapy; unless abstinence is the chosen method of contraception
* Female patients of childbearing potential must have a negative serum pregnancy test within 48 hours of transplant. Must be willing to use contraceptives from the time of study consent, during study participation, and for 16 weeks after the last dose of study agent. For sexually active men, condoms should be used during, and for at least 90 days after cessation of mycophenolate treatment. No sperm donation should be made during this period of time. For female partners of male subjects, it is recommended to use highly effective contraception during treatment and for 90 days after the last dose of mycophenolate
* No blood donation should be made by the study subjects during mycophenolate treatment and for at least 6 weeks after stopping mycophenolate treatment
* If stricter female or male contraception requirements are specified in the country-specific label for any study related therapies, they must be followed.
* Male subjects must agree to use an acceptable method for contraception for the duration of the study.

Female patients of childbearing potential must have a negative serum pregnancy test within 48 hours of transplant. Must be willing to use contraceptives from the time of study consent, during study participation, and for 16 weeks after the last dose of study agent. Reproductive Status: Definition of Women of Child-Bearing Potential (WOCBP). WOCBP comprises women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who are not post-menopausal (see definition below).

Post-menopause is defined as:

* Women who have had amenorrhea for greater than or equal to 12 consecutive months (without another cause) and who have a documented serum follicle-stimulating hormone (FSH) level > 35 mIU/mL.
* Women who have irregular menstrual periods and a documented serum FSH level > 35 mIU/mL.
* Women who are taking hormone replacement therapy (HRT).

The following women are WOCBP:

* Women using the following methods to prevent pregnancy: Oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as intrauterine devices or barrier methods (diaphragm, condoms, spermicides).
* Women who are practicing abstinence from intercourse from 2 weeks prior to administration of the 1st dose of study agent until 16 weeks after the last dose of study agent (Sexual inactivity by abstinence must be consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception)
* Women who have a partner who is sterile (e.g., due to vasectomy). WOCBP must be using an acceptable method of contraception to avoid pregnancy from the time of consent with <1% failure rate as stated in the product label throughout study participation, and for 16 weeks after the last dose of study drug in such a manner that the risk of pregnancy is minimized. Acceptable methods of contraception include: complete abstinence, any form of intra-uterine devices (without hormones), tubal sterilization or your partner has had a vasectomy.

Other acceptable forms of birth control include choosing one hormonal and one barrier method or double-barrier methods. Barrier methods include Essure®, male or female condom, diaphragm with spermicide, shield, cap with spermicide, contraceptive sponge, and spermicidals. Hormonal methods include oral contraceptive pills, transdermal patches, vaginal rings, progesterone-only, and injections. Periodic abstinence (for example, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

* These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring subjects understand how to properly use these methods of contraception.
* WOCBP must have a negative serum or urine pregnancy test result (minimum sensitivity 25 IU/L or equivalent units of HCG) within 48 hours prior to transplant (and the first dose of study drug intraoperatively).Women must not be breast-feeding

Exclusion Criteria:

* ABO incompatible donor kidney
* Deceased donor <5 years of age
* KDPI greater than or equal to 85%
* HLA identical or matched kidney
* Transplant other than kidney: has previously received a hematopoietic stem cell/marrow transplant or an organ transplant other than a kidney (with the exception of corneal transplantation)
* T- and/or B-cell positive crossmatch by complement dependent cytotoxicity or flow cytometry against the recipient
* Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria).
* Hospitalization for treatment of infection within 60 days of Day 0
* Use of parenteral (IV or IM) antibiotics (antibacterials, antivirals, anti-fungals, or anti parasitic agents) within 60 days of Day 0
* Have a history of a primary immunodeficiency
* Uncontrolled infection or any other unstable medical condition that could interfere with the study
* Seropositive for HIV, HCV or HBV, except for hepatitis B surface antibody positive
* Have a significant IgG deficiency (IgG level < 400 mg/dl) Have an IgA deficiency (IgA level < 10 mg/dL)
* Prior therapy at any time: has ever received any of the following: a) B-cell targeted therapy (e.g., rituximab, other anti-CD20 agents, anti-CD2 [epratuzumab], anti-CD52 [alemtuzumab], BLyS-receptor fusion protein [BR3], TACI fragment, crystallizable (Fc), belimumab), or IV cyclophosphamide
* Live vaccines within 30 days
* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies
* Patients with a lymphocyte count less than 500/mm3
* Patients with evidence of current drug or alcohol abuse or dependence.
* Patients with venous access limitations likely to preclude monthly infusions
* Patients whom are unlikely to comply with scheduled study visits based on investigator judgment or has a history of substance abuse, psychiatric disorder or condition that may compromise communication with the investigator
* Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiography evidence of acute ischemia or active conduction system abnormalities
* Diagnosis of liver cirrhosis or chronic viral hepatitis
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patient has received other investigational drugs within 365 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, pose a significant suicide risk
* Diagnosed or treated for malignancy within 5 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Have any other clinically significant abnormal laboratory value in the opinion of the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Foley, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospitals and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: Belimumab
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Belimumab
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 2
  40-49 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Are DSA Positive as Measured by Mean Fluorescence Intensity Greater Than Zero for DSA
Description: Use descriptive statistics to describe the rate of de novo DSA development as determined using Luminex, graft survival and function as determined by serum creatinine/eGFR and urine protein, rates of acute cellular and antibody mediated rejection.
Time Frame: 12 months from the time of transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Belimumab
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Number of Participants With DSA Development, Graft Survival, and Cellular and Antibody Rejection
Description: Use descriptive statistics to describe the rate of de novo DSA development as determined using Luminex, graft survival and function, and rates of acute cellular and antibody mediated rejection
Time Frame: 12 months from the time of transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Belimumab
Number analyzed (Participants) | 3
Participants
  DSA development | 0
  graft survival | 3
  cellular and antibody rejection | 0

3. Secondary Outcome: Report the Nature, Frequency, and Severity of Serious and Non-serious Adverse Events Greater Than or Equal to Grade 2 Per Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0.
Description: Use descriptive statistics to report the nature, frequency, and severity of serious and non-serious adverse events greater than or equal to Grade 2.
Time Frame: Monitored for 12 months from the time of transplant
Measure: Number; unit: participants
Arm/Group | Experimental: Belimumab
Number analyzed (Participants) | 3
participants
  Grade 2 : Seroma | 1
  Grade 2 : Abdominal Infection | 1
  Grade 2 : Fever | 1
  Grade 2 : Escherichia coli bacteremia from urinary tract infection | 0
  Grade 2 : Ureteral Revision | 1
  Grade 2 : Urine Leak | 1
  Grade 2 : Anaphylaxis | 1
  Grade 2 : Pseudomonas Aeruginosa Urinary Tract Infection | 1
  Grade 2 : Urinary Tract Infection | 1
  Grade 3 : Seroma | 0
  Grade 3 : Abdominal Infection | 0
  Grade 3 : Fever | 0
  Grade 3 : Escherichia coli bacteremia from urinary tract infection | 0
  Grade 3 : Ureteral Revision | 1
  Grade 3 : Urine Leak | 0
  Grade 3 : Anaphylaxis | 0
  Grade 3 : Pseudomonas Aeruginosa Urinary Tract Infection | 0
  Grade 3 : Urinary Tract Infection | 0

4. Secondary Outcome: Graft Survival and Function by Serum Creatinine
Description: Use descriptive statistics to describe the rate of graft survival and function as determined by serum creatinine
Time Frame: 1, 3, 6, 9, and 12 months from the time of transplant
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Experimental: Belimumab
Number analyzed (Participants) | 3
mg/dL
  Serum Creatinine month 1 | 3.75 [1.42 to 8.43]
  Serum Creatinine month 3 | 1.85 [1.2 to 3.01]
  Serum Creatinine month 6 | 1.57 [1.18 to 2.31]
  Serum Creatinine month 9 | 1.25 [1.08 to 1.42]
  Serum Creatinine month 12 | 1.54 [1.18 to 2.07]

5. Secondary Outcome: Graft Survival and Function by eGFR
Description: Use descriptive statistics to describe the rate of graft survival and function as determined by eGFR.
Time Frame: 1, 3, 6, 9, and 12 months from the time of transplant
Measure: Mean (Full Range); unit: mL/min/1.73m2
Arm/Group | Experimental: Belimumab
Number analyzed (Participants) | 3
mL/min/1.73m2
  eGFR month 1 | 33.33 [7 to 49]
  eGFR month 3 | 43.67 [26 to 53]
  eGFR month 6 | 49 [35 to 58]
  eGFR month 9 | 55.5 [43 to 68]
  eGFR month 12 | 48.67 [40 to 61]

6. Secondary Outcome: Graft Survival and Function by Urine Protein
Description: Use descriptive statistics to describe the rate of graft survival and function as determined by urine protein.
Time Frame: 1, 3, 6, 9, and 12 months from the time of transplant
Measure: Mean (Full Range); unit: milligrams
Arm/Group | Experimental: Belimumab
Number analyzed (Participants) | 3
milligrams
  Urine protein month 1 | 28.37 [18.3 to 44.7]
  Urine protein month 3 | 16.4 [6.8 to 31]
  Urine protein month 6 | 11.65 [6.8 to 16.5]
  Urine protein month 9 | 10 [6 to 18]
  Urine protein month 12 | 6.53 [6 to 7.6]

ADVERSE EVENTS:
Time Frame: 12 months after transplant.
Arm/Group | Experimental: Belimumab
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Belimumab (N=3)
fever (General disorders) | 1 (2)
Escherichia coli bacteremis from UTI (Infections and infestations) | 1 (1)
Ureteral Revision (Injury, poisoning and procedural complications) | 1 (1)
Urine Leak (Renal and urinary disorders) | 1 (1)
Klebsiella Pneumoniae UTI (Infections and infestations) | 1 (1)
Pseudomonas Aeruginosa UTI (Infections and infestations) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Subtotal Parathyroidectomy (Renal and urinary disorders) | 1 (1)
Post-surgical fluid collection (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Belimumab (N=3)
Urinary Tract Infection (Infections and infestations) | 1 (1)
tremors (Nervous system disorders) | 1 (1)
Elevated Donor Specific Antibody (General disorders) | 1 (1)
Forgetfulness (General disorders) | 1 (1)
Night Sweats (General disorders) | 1 (1)
Generalized Edema (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (2)
Chills (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Right distal fibula fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (3)
Glucosuria (Renal and urinary disorders) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 1 (1)
Delayed Graft Function (Renal and urinary disorders) | 1 (1)
Bladder Spasms (Renal and urinary disorders) | 1 (1)
Urine Leak (Renal and urinary disorders) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seroma (Surgical and medical procedures) | 1 (1)
Right Genitofemoral Neuralgia (Surgical and medical procedures) | 1 (1)
Post operative pain at drain site (Surgical and medical procedures) | 1 (1)
Cytomegalovirus (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT03591380/Prot_SAP_000.pdf